CLINICAL TRIAL: NCT06863012
Title: EUS-guided Portal Pressure Gradient (PPG) Measurement: a Potential Alternative to the Traditional HVPG
Acronym: EUS-PPG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio Privada Mon Clinic Barcelona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EUS-PPG
Record Dates: First submitted 2025-02-25; First posted 2025-03-07 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Portal Hypertension; Chronic Liver Disease (CLD); Cirrhosis
Keywords: Hepatic Venous Pressure Gradient; Endoscopic Ultrasound-Guided Portal Pressure Gradient; Portal hypertension; Non-Invasive Diagnostic Methods for Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EUS-PPG and HVPG Measurement in Portal Hypertension (Experimental)
  Interventions: Diagnostic Test: Endoscopic Ultrasound-Guided Portal Pressure Gradient (EUS-PPG) Measurement; Diagnostic Test: Hepatic Venous Pressure Gradient (HVPG) Measurement

INTERVENTIONS:
Diagnostic Test: Endoscopic Ultrasound-Guided Portal Pressure Gradient (EUS-PPG) Measurement — Endoscopic Ultrasound-Guided Portal Pressure Gradient (EUS-PPG) measurement is a minimally invasive, ultrasound-based diagnostic procedure designed to assess portal hypertension in patients with chronic liver disease. Using an endoscopic ultrasound (EUS) probe, and a fine-needle aspiration (FNA) needle (EchoTip® Insight™) is used to directly measure intravascular pressures. Unlike the standard hepatic venous pressure gradient (HVPG) measurement, EUS-PPG provides direct pressure readings, does not require catheterization of the hepatic vein, and eliminates the need for radiation, iodinated contrast, and interventional radiology. This study aims to evaluate the accuracy, feasibility, and safety of EUS-PPG compared to HVPG.
Diagnostic Test: Hepatic Venous Pressure Gradient (HVPG) Measurement — Hepatic Venous Pressure Gradient (HVPG) measurement is the current gold standard for assessing portal hypertension in patients with chronic liver disease. The procedure involves catheterization of the hepatic vein via the jugular or femoral vein, where free hepatic venous pressure (FHVP) and wedged hepatic venous pressure (WHVP) are measured using a pressure transducer. HVPG is an indirect measure of portal pressure and requires fluoroscopy, radiation exposure, and specialized interventional radiology equipment. While widely used in clinical practice, HVPG has limitations, including the need for a hospital setting, potential patient discomfort, and limited feasibility in certain cases. This study will compare HVPG to EUS-PPG to determine whether EUS-PPG can serve as a less invasive and more accessible alternative.

SUMMARY:
The goal of this investigator-initiated, single-arm, prospective study is to evaluate the accuracy, safety, and feasibility of endoscopic ultrasound-guided portal pressure gradient (EUS-PPG) measurement as a potential alternative to the traditional hepatic venous pressure gradient (HVPG) method in patients with portal hypertension due to chronic liver disease. The main questions it aims to answer are:

* What is the correlation between EUS-PPG and HVPG measurements in patients with portal hypertension due to cirrhosis?
* Can EUS-PPG serve as a reliable and less invasive alternative to HVPG for assessing portal pressure?
* What are the safety outcomes associated with EUS-PPG compared to HVPG?

Researchers will compare EUS-PPG measurements with HVPG measurements within the same patients to assess whether EUS-PPG provides accurate and clinically comparable portal pressure readings while reducing procedural risks.

Participants will:

* Be adults aged 18 to 85 with a history of liver disease and portal hypertension or suspected cirrhosis requiring HVPG measurement.
* Undergo both EUS-PPG and HVPG measurements within a seven-day window to allow for direct comparison of results.
* Receive standard clinical care for their condition, including routine diagnostic evaluations and portal hypertension management as needed.
* Be monitored for safety outcomes, including adverse events such as bleeding, infection, perforation, and any other complications related to the procedure.
* Provide relevant demographic and clinical data, including liver disease history, Child-Pugh and MELD scores, and portal hypertension-related complications such as varices or ascites.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 to 85 years of age inclusive, at the time of signing the informed consent form.
* Subjects who have a history of liver disease and portal hypertension or suspected cirrhosis requiring HVPG measurement.
* Subjects capable of giving signed informed consent.

Exclusion Criteria:

* Pregnancy.
* Significant bleeding risk (International Normalized Ratio (INR) > 1.5 OR platelet count < 50000).
* Presence of active gastrointestinal bleeding at the time of screening
* History of any blood thinner consumption (e.g. warfarin, heparin, novel roal anticoagulants) within the last 5 days.
* Presence of massive ascites causing abdominal distension or requiring frequent therapeutic paracentesis.
* Subjects having received previous Transjugular Intrahepatic Portosystemic Shunt (TIPS) or Surgical Portosystemic Shunt.
* Hepatocellular carcinoma not meeting Milan Criteria.
* Presence of portal vein thrombosis or another suspected component of presinusoidal portal hypertension.
* Presence of extra-hepatic cancer, terminal disease, or severe comorbidities significantly limiting life expectancy or affecting study participation.
* Stenosis or surgical anatomical alterations of the gastrointestinal tract that could preclude endoscopic access with the echoendoscope.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between the portosystemic pressure gradient (PPG) measured directly via endoscopic ultrasonography (EUS-PPG) and measured via the hepatic venous pressure gradient (HVPG). | 7 days
  Correlation between the portosystemic pressure gradient (PPG) measured directly via endoscopic ultrasonography (EUS-PPG) using the EchoTip® Insight™ needle and the hepatic venous pressure gradient (HVPG) measured through hepatic vein catheterization in patients with chronic portal hypertension due to liver cirrhosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Barcelona, Spain